CLINICAL TRIAL: NCT03811743
Title: A Coordinated Parent/Child Dyad Weight Loss Intervention: Dyad Plus (Feasibility)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055004
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2021-05

CONDITIONS: Weight Loss; Pediatric Obesity
Keywords: Youth; Parents; Overweight; Families
MeSH Terms: conditions — Weight Loss; Pediatric Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents Participants (Experimental): Adolescents will participate in the Dyad Plus program along with their caregivers. The Dyad plus program consist of the combination of two existing programs (Brenner FIT for adolescents and By Design for the adult caregivers) with a new, novel coordination component
  Interventions: Behavioral: Brenner FIT; Behavioral: Coordination
- Caregivers of adolescents participants (Experimental): Adult caregivers will participate in the Dyad Plus program along with their youth participants. The Dyad plus program consist of the combination of two existing programs (Brenner FIT for adolescents and By Design for the adult caregivers) with a new, novel coordination component
  Interventions: Behavioral: By Design; Behavioral: Coordination

INTERVENTIONS:
Behavioral: Brenner FIT — Brenner FIT pediatric weight management program enrollment. an interdisciplinary, family-based pediatric weight management clinic based upon the Familial Approach to Treatment of Childhood Obesity. Patients are referred by a physician for obesity or overweight with a weight-related comorbidity. Treatment teams are comprised of a pediatrician, counselor, dietitian, and physical activity specialist, with others (e.g., social workers, physical therapists) as needed. The entire family is encouraged to attend all aspects of the treatment program, although only one attending caregiver is required.
  Arms: Adolescents Participants
Behavioral: By Design — Weight loss program for adults/caregivers of those enrolled in Brenner FIT. Participants in the By Design condition (adult caregivers) will be prescribed the Essentials lifestyle intervention which includes tailored dietary and physical activity goals designed to achieve 1-2 lbs./week of weight loss, provided by a multidisciplinary team of medical providers, dietitians, behaviorists, and exercise specialists. A daily calorie restriction of 500 kcal/day is prescribed based on estimates of total energy expenditure (TEE) obtained from a measured resting metabolic rate (RMR) prior to enrollment.
  Arms: Caregivers of adolescents participants
Behavioral: Coordination — This component adds four additional strategies: dyad group sessions, one-on-one parent/child communication sessions, joint goal setting/tracking, and home environment assessment. This innovative approach will seek to employ components of motivation and communication theories to increase self-monitoring, positive communication, problem solving, and social support to increase healthy physical activity and eating behaviors to increase the effectiveness of the weight loss programs beyond gains observed in matched controls.
  Essentials (adults), with four additional components: dyad group sessions, one-on-one parent/child communication sessions, joint goal setting/tracking, and home environment assessment

SUMMARY:
The purpose of this research is to develop a coordinated program (Dyad Plus) that would help to facilitate self-monitoring, positive communication, joint problem solving, and social support to increase physical activity, healthy eating, and weight loss. Participants of the Brenner FIT (Families In Training) pediatric weight management program and their parent/guardian will co-enroll in weight loss programs. Parents/guardians will receive the components of By Design Essentials.

DETAILED DESCRIPTION:
Participation in this study will involve participation in six, one-hour sessions in addition to those required by your weight loss program. These sessions will work to facilitate an increase in self-monitoring, positive communication, problem solving, and social support to increase healthy physical activity and eating behaviors to increase the effectiveness of the weight loss programs. Joint goal setting and tracking will be enabled by commercially available devices and apps. Each caregiver and child will receive an activity monitor, activity app, and a food app (digital food diary) that allows self-monitoring of consumption and "social accountability," which will allow caregivers and the Brenner FIT team to monitor and encourage. Furthermore, two home visits will be conducted to evaluation the home food and activity environments to inform tailored feedback to families.

Brenner FIT is a family-based pediatric weight management clinic for youth 2-18 years old referred by a physician for overweight or obesity.11-14 By Design is an adult (>18yrs) weight loss clinic that includes tailored dietary and physical activity behavioral counseling. The preliminary data suggest that most adolescent youth who enroll in Brenner FIT have at least one adult caregiver who is eligible and would benefit from enrollment in By Design Essentials.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for enrollment in Brenner FIT and/or By Design Essentials
* Caregiver who lives in the house with a BMI > 30
* No contraindication for physical activity or caloric restriction
* Must be able to read and write English

Exclusion Criteria:

* Over the age of 65
* BMI < 30
* Contraindication for physical activity or caloric restriction
* Cannot read or write English

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
BMI z-score | Baseline
  Weight status of caregivers and youth will be quantified through calculation of BMI derived from measurement of height and weight at the intake and follow-up visits. Both height (plus or minus 0.1 cm) and weight (plus or minus 0.5 kg) will be recorded twice and values will be averaged to produce the final value using a Tanita (registered trademark) digital scale and a Seca (registered trademark) Height Rod (respectively). BMI will be calculated as kg /m2. BMI z-score will be calculated using CDC growth charts.
BMI z-score | 3 Months
  Weight status of caregivers and youth will be quantified through calculation of BMI derived from measurement of height and weight at the intake and follow-up visits. Both height (plus or minus 0.1 cm) and weight (plus or minus 0.5 kg) will be recorded twice and values will be averaged to produce the final value using a Tanita (registered trademark) digital scale and a Seca (registered trademark) Height Rod (respectively). BMI will be calculated as kg /m2. BMI z-score will be calculated using CDC growth charts.
BMI z-score | 6 months
  Weight status of caregivers and youth will be quantified through calculation of BMI derived from measurement of height and weight at the intake and follow-up visits. Both height (plus or minus 0.1 cm) and weight (plus or minus 0.5 kg) will be recorded twice and values will be averaged to produce the final value using a Tanita (registered trademark) digital scale and a Seca (registered trademark) Height Rod (respectively). BMI will be calculated as kg /m2. BMI z-score will be calculated using CDC growth charts.

SECONDARY OUTCOMES:
Physical Activity Assessed by Accelerometry | Baseline
  Physical activity data will be collected using ActiGraph (trademark) accelerometers worn continuously over 7 days except during bathing and sleeping. Moderate to vigorous activity will be measured in minutes.
Physical Activity Assessed by Accelerometry | 6 months
  Physical activity data will be collected using ActiGraph (trademark) accelerometers worn continuously over 7 days except during bathing and sleeping. Moderate to vigorous activity will be measured in minutes.
Physical Activity Assessed by PAQ-A | Baseline
  The Physical Activity Questionnaire for Adolescents (PAQ-A) will be given to assess physical activity.
  The PAQ-A ranges from 1-7. Higher score denotes better outcome.
Physical Activity Assessed by PAQ-A | 6 months
  The Physical Activity Questionnaire for Adolescents (PAQ-A) will be given to assess physical activity.
  The PAQ-A ranges from 1-7. Higher score denotes better outcome.
Physical Activity Assessed by IPAQ | Baseline
  The International Physical Activity Questionnaire (IPAQ) will be given to assess physical activity in adults.
  The IPAQ ranges from 10-960 minutes/day of physical activity. Higher score denotes better outcome.
Physical Activity Assessed by IPAQ | 6 months
  The International Physical Activity Questionnaire (IPAQ) will be given to assess physical activity in adults.
  The IPAQ ranges from 10-960 minutes/day of physical activity. Higher score denotes better outcome.
Caloric intake expressed in kcals | Baseline
  Diet will be assessed by the Automated Self-Administered 24-hour (ASA24) dietary assessment tool.
Caloric intake expressed in kcals | 6 months
  Diet will be assessed by the Automated Self-Administered 24-hour (ASA24) dietary assessment tool.
Concentration of fasting glucose for all participants, mg/dL | Baseline
  Fasting blood glucose will be ascertained for each participant. A fasting blood sugar level less than 100 mg/dL (5.6 mmol/L) is optimal. A fasting blood sugar level from 100 to 125 mg/dL (5.6 to 6.9 mmol/L) is considered prediabetes.
Concentration of fasting glucose for all participants, mg/dL | 6 months
  Fasting blood glucose will be ascertained for each participant. A fasting blood sugar level less than 100 mg/dL (5.6 mmol/L) is optimal. A fasting blood sugar level from 100 to 125 mg/dL (5.6 to 6.9 mmol/L) is considered prediabetes.
Concentration of fasting Insulin for all participants, mg/dL | Baseline
  Fasting insulin levels will be gathered from all participants.
Concentration of fasting Insulin for all participants, mg/dL | 6 months
  Fasting insulin levels will be gathered from all participants.
Hemoglobin A1c concentration for all participants, measured in percentage | Baseline
  Normal range for the hemoglobin A1c level is between 4% and 5.6%. Hemoglobin A1c levels between 5.7% and 6.4% Values greater denote diabetes.
Hemoglobin A1c concentration for all participants, measured in percentage | 6 months
  Normal range for the hemoglobin A1c level is between 4% and 5.6%. Hemoglobin A1c levels between 5.7% and 6.4%. Values greater denote diabetes.
Aspartate Aminotransferase -Levels of AST for all participants, measured in units per liter (IU/L) | Baseline
  AST a useful test for detecting or monitoring liver damage.
Aspartate Aminotransferase -Levels of AST for all participants, measured in units per liter (IU/L) | 6 months
  AST a useful test for detecting or monitoring liver damage.
Alanine Aminotransferase-Levels of ALT for all participants, measured in units per liter | Baseline
  A low level of ALT in the blood is expected and is normal.
Alanine Aminotransferase-Levels of ALT for all participants, measured in units per liter | 6 months
  A low level of ALT in the blood is expected and is normal.
Concentration of total cholesterol (mg/dL) | Baseline
  total cholesterol: less than 200 mg/dL
Concentration of total cholesterol (mg/dL) | 6 months
  total cholesterol: less than 200 mg/dL
Economic costs of the three intervention arms over duration of program (USD) | Baseline through 6 months
  Clinical and non-clinical costs of the interventions will be compiled over the duration of the program. All cost will be reported in the same unit.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Moore, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skelton JA, Beech BM. Attrition in paediatric weight management: a review of the literature and new directions. Obes Rev. 2011 May;12(5):e273-81. doi: 10.1111/j.1467-789X.2010.00803.x. Epub 2010 Sep 29. PMID 20880126

DOCUMENTS (1):
  • Informed Consent Form (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03811743/ICF_000.pdf